CLINICAL TRIAL: NCT03958110
Title: Analysis of the Variation in Thickness of Per-papillary Retinal Optic Nerve Fibres in Professional Rugby Players
Acronym: ON RUGBY
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMT_2019_3
Record Dates: First submitted 2019-05-20; First posted 2019-05-21 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Rugby Professionals; Concussion
Keywords: Retinophotography; OCT; Optical nerve
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: OCT A — OCT (Optical Coherence Tomography) and Retinophotography made at the beginning and end of the Rugby season.

SUMMARY:
The main hypothesis is that exposure to repeated shocks is associated with a greater decrease in the thickness of optical nerve fibres.

In order to show a association between the occurrence of concussions (in number and severity) and the variation in the thickness of the retinal nerve fibre layer, all participating rugby players will have an ophthalmologic examination (OCT and (retinophotography) at the beginning and end of the Rugby season.

ELIGIBILITY:
Inclusion Criteria:

* Professional rugby player

Exclusion Criteria:

* impossibility to realise OCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Professional rugby players
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Average thickness difference of the RNFL on each eye in micrometers measured by OCT, between the beginning and the end of the season | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Opthalmologique A de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No